CLINICAL TRIAL: NCT01162811
Title: Visualization and Structured Attention Behaviour -- Does it Reduce the Patient's Experience of Pain Intensity and Anxiety During Ablation of Atrial Fibrillation?
Brief Title: Visualization and Structured Attention Behaviour for Pain and Anxiety Reduction During Ablation of Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Marianne Wetendorff Noergaard, Cardiac Cath.lab 2012, Rigshospitalet. Blegdamsvej 9, DK- 2100, Copenhagen Ø Denmark
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: J. nr. 2007-58-0015.).
Record Dates: First submitted 2010-07-08; First posted 2010-07-15 (Estimated); Last update posted 2011-07-21 (Estimated); Status verified 2009-11

CONDITIONS: Atrial Fibrillation
Keywords: Visualization; relaxation; self hypnotic relaxation; hypnosis; invasive medical procedures; atrial fibrillation; ablation; catheter ablation; pain; anxiety
MeSH Terms: conditions — Atrial Fibrillation; Pain; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention): The control group receives conventional care and treatment
- Intervention group (Experimental): the intervention group receives visualization and relaxation exercises together with structured behavioural attention
  Interventions: Behavioral: visualization together with structured behavioural attention.

INTERVENTIONS:
Behavioral: visualization together with structured behavioural attention. — visualization and relaxation exercises together with structured behavioural attention.
  Arms: Intervention group

SUMMARY:
The purpose of this study is to test the efficacy of visualization and relaxation exercises together with a structured behavioural attention from nurses during ablation of atrial fibrillation.

The study will test the following hypothesis which is also aim for intervention:

Relaxation and visualization performed in patients during ablation of atrial fibrillation combined with structured attention behaviour from the nurse reduces the patient's experience of pain and anxiety - and secondary reduces the consumption of painkillers and the number of episodes of adverse outcome that requires extra attention from staff.

The survey is conducted as a controlled trial with a control group and an intervention group.

DETAILED DESCRIPTION:
Background:

Atrial fibrillation (AF) is the most common form of cardiac arrhythmia with a prevalence of 5% among people older than 65 years, and 0.4% of the total population. Ablation is a relatively new treatment that has proven to be effective in removing physical symptoms in patients with severe symptoms.

Compared to other ablation treatments, ablation of AF is complex and of longer duration. It can be accompanied by significant discomfort and pain, despite pharmacological analgesia.

Non pharmacological analgesia in the form of relaxation exercises and visualization has successfully been used to reduce the experience of pain intensity and anxiety of other invasive procedures.

Aim:

The study will test the following hypothesis which also acts as aim for intervention:

Relaxation and visualization performed in patients during ablation of atrial fibrillation combined with structured attention behaviour from the nurse reduces the patient's experience of pain and anxiety - and secondary reduces the consumption of painkillers and the number of episodes of adverse outcome that requires extra attention from staff.

Design / Methodology:

The Trial is conducted in a cardiac lab. The survey is conducted as a controlled Trial. The control group receives conventional care and treatment and the intervention group receives visualization and relaxation exercises together with structured behavioural attention.

The patient scores experienced pain intensity and anxiety in a validated linear numerical rank scale.

A Statistical calculation of power estimated the required number of patients to 70 in each group.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for ablation of atrial fibrillation

Exclusion Criteria:

* Unable to give informed consent
* Impaired mental function, psychosis, severe chronic obstructive pulmonary disease, intolerance towards midazolam or fentanyl
* Undergoing the ablation in general anaesthesia
* Unable to speak or understand danish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2009-11; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Pain and anxiety is determined from self-reporting by the patient on a validated NRS scale. | Day 1 :Patient self-reporting every 15 minutes from the onset of the ablation procedure to the end of the ablation procedure. In addition self-reporting is recorded if the patient complains in between these fixed measurement points. No follow-up.

SECONDARY OUTCOMES:
Amount of Medication used /kg (Fentanyl and Midazolam) during the ablation procedure) | Day 1: From the onset to the end of the ablation procedure. No follow-up.
Number of adverse events during the ablation procedure | Day 1: Are recorded whenever they occur from the onset, to the end of the ablation procedure. No follow-up.
  Defined as occurrences requiring extra medical attention to restore hemodynamic and cardiorespiratory stability during the procedure, including systolic blood pressure fluctuation, vasovagal episodes, cardiac events and respiratory impairment

CONTACTS AND LOCATIONS:
Overall Officials: Preben U Pedersen, RN, PhD, Study Chair — The Cardiac Cath.lab. The Heartcenter,Rigshospitalet, Copenhagen Denmark
Locations (1):
- Coepenhagen University Hospital, Rigshospitalet, Copenhagen, Copenhagen Ø, Denmark